CLINICAL TRIAL: NCT00406913
Title: Assessment of Conjunctival Flora and Optimal Ocular Sterilization Technique Prior to Cataract Surgery Using Intranasal Mupirocin Ointment
Brief Title: Prophylaxis Prior to Cataract Surgery Conjunctival Flora and Optimal Ocular Sterilization Technique Prior to Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14208B
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Endophthalmitis; Cataract Surgery; Prophylaxis
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Mupirocin ointment (Experimental)
  Interventions: Drug: mupirocin ointment; Other: SOC sterilization
- Standard of Care sterilization (Active Comparator)
  Interventions: Other: SOC sterilization

INTERVENTIONS:
Drug: mupirocin ointment
  Arms: Mupirocin ointment
Other: SOC sterilization

SUMMARY:
The purpose of this study is to evaluate the conjunctival flora prior to cataract or vitrectomy surgery comparing mupirocin ointment applied to the conjunctiva along with standard ocular sterilization vs. standard ocular sterilization alone.

DETAILED DESCRIPTION:
Bacterial endophthalmitis is a rare but devastating complication of intraocular surgery. Given the devastating ocular sequelae of endophthalmitis, one cannot underestimate the need to develop a sterilization strategy which most effectively prevents intraocular infection. The most common organisms causing bacterial postoperative endophthalmitis are gram-positive cocci, particularly coagulase-negative staphylococci and Staphylococcus Aureus. It is thought that the most common sources of bacterial contamination predisposing to endophthalmitis are the eyelids and conjunctiva (Ariyasu).

The two main techniques used to reduce the bacterial flora on the ocular surface include treatment of the ocular surface with topical antibiotics prior to surgery and the instillation of 5% povidone-iodine during the prep immediately prior to beginning the surgical procedure (Speaker). Mupirocin ointment is a logical choice for surgical prophylaxis as it has been reported that mupirocin treatment applied to the nose resulted in elimination rates (of S. Aureus from the nares) of 91% directly after therapy (Doebbeling). Use of mupirocin ointment applied to the nares prior to eye surgery resulted in a significant decrease in the bacterial load on the conjunctiva at the time of surgery (Alexandrou, in press). Using mupirocin ointment directly to the conjunctiva, in addition to standard ocular sterilization techniques, may result in an even greater decrease in conjunctival flora prior to eye surgery.

ELIGIBILITY:
Inclusion Criteria:

* Included in the study will be any patient eligible for cataract or vitrectomy surgery. No populations will be excluded on the basis of demographics.

Exclusion Criteria:

* Excluded will be those patients who have known sensitivity or allergy to mupirocin ointment, or patients using topical ocular or systemic antibiotics during a two week period prior to entry into the study. Additionally, patient's using topical corticosteroids will be excluded as well

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Positive conjunctival culture | pre and post op

CONTACTS AND LOCATIONS:
Overall Officials: Seenu Hariprasad, MD, Principal Investigator — University of Chicago Hospitals
Locations (1):
- University of Chicago Hospitals, Chicago, Illinois, United States

REFERENCES:
- [Background] Speaker MG, Menikoff JA. Prophylaxis of endophthalmitis with topical povidone-iodine. Ophthalmology. 1991 Dec;98(12):1769-75. doi: 10.1016/s0161-6420(91)32052-9. PMID 1775308
- [Background] Kluytmans JA, Wertheim HF. Nasal carriage of Staphylococcus aureus and prevention of nosocomial infections. Infection. 2005 Feb;33(1):3-8. doi: 10.1007/s15010-005-4012-9. PMID 15750752
- [Background] Ariyasu RG, Nakamura T, Trousdale MD, Smith RE. Intraoperative bacterial contamination of the aqueous humor. Ophthalmic Surg. 1993 Jun;24(6):367-73; discussion 373-4. PMID 8336886
- [Background] Doebbeling BN, Breneman DL, Neu HC, Aly R, Yangco BG, Holley HP Jr, Marsh RJ, Pfaller MA, McGowan JE Jr, Scully BE, et al. Elimination of Staphylococcus aureus nasal carriage in health care workers: analysis of six clinical trials with calcium mupirocin ointment. The Mupirocin Collaborative Study Group. Clin Infect Dis. 1993 Sep;17(3):466-74. doi: 10.1093/clinids/17.3.466. PMID 8218691